CLINICAL TRIAL: NCT05007951
Title: A 2-Stage, Phase III, Randomized, Active-controlled, Observer-blind, Parallel-group, Multi-center Study to Assess the Immunogenicity and Safety of SK SARS-CoV-2 Recombinant Nanoparticle Vaccine Adjuvanted With AS03 (GBP510) in Adults Aged 18 Years and Older
Brief Title: Immunogenicity and Safety Study of SK SARS-CoV-2 Recombinant Nanoparticle Vaccine (GBP510) Adjuvanted With AS03 (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Collaborators: International Vaccine Institute (Other); GlaxoSmithKline (Industry); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GBP510_003
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome assessors are unblinded after Stage1 interim analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Test group (GBP510) - Cohort 1 (Experimental): Immunogenicity Cohort
  Interventions: Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose)
- Control group (ChAdOx1-S) - Cohort 1 (Active Comparator): Immunogenicity Cohort
  Interventions: Biological: ChAdOx1-S not less than 2.5 × 10^8 infectious units
- Test group (GBP510) - Cohort 2 (Experimental): Safety Cohort
  Interventions: Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose)
- Control group (ChAdOx1-S) - Cohort 2 (Active Comparator): Safety Cohort
  Interventions: Biological: ChAdOx1-S not less than 2.5 × 10^8 infectious units
- Test group (GBP510) - Cohort 3 (Experimental): Booster Subcohort
  Interventions: Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose)
- Control group (ChAdOx1-S) - Cohort 3 (Active Comparator): Booster Subcohort
  Interventions: Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose)

INTERVENTIONS:
Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose) — injection volume of 0.5mL on days 0 and 28 (stage1)
  Arms: Test group (GBP510) - Cohort 1; Test group (GBP510) - Cohort 2
Biological: ChAdOx1-S not less than 2.5 × 10^8 infectious units — injection volume of 0.5mL on days 0 and 28 (stage1)
  Arms: Control group (ChAdOx1-S) - Cohort 1; Control group (ChAdOx1-S) - Cohort 2
Biological: GBP510 adjuvanted with AS03 (Receptor-Binding Domain(RBD) 25ug/dose) — injection volume of 0.5mL on days 0 (stage2)
  Arms: Control group (ChAdOx1-S) - Cohort 3; Test group (GBP510) - Cohort 3

SUMMARY:
This is a 2-Stage, Phase III, randomized, active-controlled, observer-blind, parallel-group, multi-center study to compare the immunogenicity and safety of SK SARS-CoV-2 recombinant nanoparticle vaccine adjuvanted with AS03 (GBP510) to ChAdOx1-S in adults aged 18 years and older.

DETAILED DESCRIPTION:
The purpose of this study is to assess the immunogenicity and safety of SK SARS-CoV-2 recombinant nanoparticle vaccine adjuvanted with AS03 (GBP510) in adults aged 18 years and older.

This study includes 2-dose schedule (28-day interval) of GBP510(Test vaccine) and ChAdOx1-S(Control vaccine) in stage1. Participants are expected to participate for up to a maximum of approximately 13 months. A 12-month study follow-up after the 2nd vaccination will be conducted. One booster dose of GBP510 is scheduled for both test group and control group in Stage2. A 12-month study follow-up after the 3rd vaccination will be conducted.

International Vaccine Institute (IVI) conducts GBP510_003 trial as co-sponsor with SK bioscience.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age and older, at the time of signing the informed consent;
* Participants who are healthy or medically stable as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, and medical judgement of the investigator;
* Participants who are able to attend all scheduled visits and comply with all study procedures;
* Female participants of childbearing potential must agree to be heterosexually inactive, or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the 1st study vaccination to 12 weeks after the last study vaccination;
* Female participants with a negative urine or serum pregnancy test at screening;
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in protocol;

<Stage2>

* Participants who have received 2 doses of GBP510 25μg adjuvanted with AS03 or ChAdOx1-S and have blood samples until Visit 7 in Stage 1
* Participants who received a primary series of GBP510 or ChAdOx1-S at least 12 weeks prior to booster vaccination in Stage 2
* Participants who are able to attend all additionally scheduled visits and comply with all study procedures.
* Female participants of childbearing potential must agree to be heterosexually inactive, or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the booster dose (3rd study vaccination) to 12 weeks after the booster dose
* Female participants with a negative urine or serum pregnancy test prior to the booster dose (the third dose of study vaccine)
* Capable of giving an informed consent for Stage 2 study in compliance with the requirements and restrictions listed in the informed consent form (ICF) for Stage 2 and in this protocol.

Exclusion Criteria:

* Any clinically significant respiratory symptoms (e.g., cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 72 hours prior to the 1st study vaccination. A prospective participant should not be included until 72 hours after the condition has resolved;
* (Only for Cohort 1) Prior SARS-CoV-2 infection or vaccination confirmed by a positive result of qualitative test for SARS-CoV-2 antibody using a rapid antibody kit at screening;
* History of virologically-confirmed SARS or MERS disease, or SARS / MERS vaccination;
* History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease;
* History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination;
* History of hypersensitivity and severe allergic reaction (e.g., anaphylaxis, Guillain-Barre syndrome) to any vaccines or components of the study vaccine;
* History of malignancy within 1 year prior to the 1st study vaccination (with the exception of malignancy with minimal risk of recurrence at the discretion of the investigator);
* Significant unstable chronic or acute illness that, in the opinion of the investigator, might pose a health risk to the participant if enrolled, or could interfere with the protocol-specified activities, or interpretation of study results;
* Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions);
* Female participants who are pregnant or breastfeeding;
* Receipt of any vaccine within 4 weeks prior to the 1st study vaccination or planned receipt of any vaccine from enrollment through 28 days after the last study vaccination (Visit 7), except for influenza vaccination, which may be received at least 2 weeks prior to the 1st study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines;
* Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the 1st study vaccination;
* Receipt of any medications or vaccinations intended to prevent COVID-19;
* Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anticancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the 1st vaccination. The use of topical and nasal glucocorticoids will be permitted;
* Participation in another clinical study involving study intervention within 4 weeks prior to the 1st study vaccination, or concurrent, planned participation in another clinical study with study intervention during the study period.
* Participants who are subjected to any global or local restrictions in place for use of ChAdOx1-S (e.g. age, gender, or other specific population groups)
* Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.

<Stage2>

* Any clinically significant respiratory symptoms (e.g., cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 72 hours prior to the booster dose (3rd study vaccination). A prospective participant should not be included until 72 hours after the condition has resolved.
* History of confirmed COVID-19, SARS or MERS disease confirmed by serological, virological assay, or rapid antigen kit
* Receipt of any medications or vaccinations intended to prevent COVID-19 except for GBP510 or ChAdOx1-S.
* Receipt of any vaccine within 4 weeks prior to the booster vaccination or planned receipt of any vaccine from enrollment through 28 days after the booster vaccination (Visit 4B), except for influenza vaccination, which may be received at least 2 weeks prior to the booster vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the booster vaccination
* Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the booster vaccination. The use of topical and nasal glucocorticoids will be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4036 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer(GMT) of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays | 2 weeks post 2nd vaccination
  For Cohort 1
Percentage of participants with ≥ 4-fold rise in wild-type virus neutralizing antibody titer from baseline | 2 weeks post 2nd vaccination
  For Cohort 1
Geometric Mean Titer(GMT) of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays | 2 weeks post 3rd (booster) and 2nd vaccination
  For Cohort 3

SECONDARY OUTCOMES:
GMT of SARS-CoV-2 Receptor-Binding Domain(RBD)-binding IgG antibody measured by Enzyme-Linked Immunosorbent Assay (ELISA) at each time point post-vaccination | Through Day 365 post last vaccination
  For Cohort 1
Geometric Mean Fold Rise(GMFR) of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA from baseline | Through Day 365 post last vaccination
  For Cohort 1
Percentage of participants with ≥ 4-fold rise SARS-CoV-2 RBD-binding IgG titer from baseline | Through Day 365 post last vaccination
  For Cohort 1
GMT of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays | Through Day 365 post last vaccination
  For Cohort 1
GMFR of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays from baseline | Through Day 365 post last vaccination
  For Cohort 1
Percentage of participants with ≥ 4-fold rise in wild-type virus neutralizing antibody titer from baseline | Through Day 365 post last vaccination
  For Cohort 1
Cell-mediated response for both Th1 and Th2 cytokines measured by Enzyme-Linked ImmunoSpot (ELISpot)/ FluoroSpot, and for both CD4+ and CD8+ T-cells measured by Fluorescence-activated cell sorting(FACS) | Through Day 365 post last vaccination
  For Cohort 1
Occurrence of immediate systemic reactions in the 30 minutes post each vaccination | Through 30 minutes post each vaccination
  For all Cohort
Occurrence of solicited local Adverse Events(AEs) | Through 7 days post each vaccination
  For all Cohort
Occurrence of solicited systemic AEs | Through 7 days post each vaccination
  For all Cohort
Occurrence of unsolicited AEs | Through 28 days post each vaccination
  For all Cohort
Occurrence of Serious Adverse events(SAEs), Medically attended Adverse Events(MAAEs), AEs leading to study withdrawal, and Adverse Events of Special Interests(AESIs) | Through Day 365 post last vaccination
  For all Cohort
GMTs of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays | 2 weeks post 3rd (booster) and 2nd vaccination
  For Cohort 3
Percentages of participants with ≥ 4-fold rise in wild-type virus neutralizing antibody titer from baseline (Visit 2) | 2 weeks post 3rd (booster) and 2nd vaccination
  For Cohort 3
GMTs of neutralizing antibody to the SARS-CoV-2 measured by wild-type virus neutralization assays | pre (Visit 1B) and 2 weeks post 3rd (booster) vaccination
  For Cohort 3
GMTs of neutralizing antibody to the SARS-CoV-2 measured by neutralization assays | 2 weeks post 3rd (booster) and 2nd vaccination
  For Cohort 3
GMT of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA at each time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
GMFR of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA from baseline (Visit 2) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
GMFR of SARS-CoV-2 RBD-binding IgG antibody measured by ELISA from prior to booster vaccination (Visit 1B) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
Percentage of participants with ≥4-fold rise in ELISA SARS-CoV-2 RBD-binding IgG titer from baseline (Visit 2) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
Percentage of participants with ≥4-fold rise in ELISA SARS-CoV-2 RBD-binding IgG titer from pre-booster vaccination (Visit 1B) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
GMT of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay at each time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
GMFR of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay from baseline (Visit 2) to each subsequent time point post booster vaccination. | Through Day 365 post last vaccination
  For Cohort 3
GMFR of neutralizing antibody to SARS-CoV-2 measured by wild-type virus neutralization assay from prior to booster vaccination (Visit 1B) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
Percentage of participants with ≥4-fold rise in wild-type virus neutralizing antibody titer to SARS-CoV-2 from baseline (Visit 2) to each subsequent time point post booster vaccination. | Through Day 365 post last vaccination
  For Cohort 3
Percentage of participants with ≥4-fold rise in wild-type virus neutralizing antibody titer to SARS-CoV-2 from pre-booster vaccination (Visit 1B) to each subsequent time point post booster vaccination | Through Day 365 post last vaccination
  For Cohort 3
Cell-mediated response for both Th1 and Th2 cytokines (including but not limited to INF-γ, TNF-α, IL-2, and IL-4 produced by T lymphocytes) measured by ELISpot and/or FluoroSpot, and for both CD4+ and CD8+ T-cells measured by FACS | Through Day 365 post last vaccination
  For Cohort 3

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, Principal Investigator — Korea University Guro Hospital
Locations (38):
- New Zealand (7):
  - Southern Clinicaltrials Waitemata, Auckland
  - Southern Clinical Trials Christchurch, Christchurch
  - Lakeland Clinicaltrials Waikato, Hamilton
  - Southern Clinical Trials Tasman, Nelson
  - Lakeland Clinicaltrials Culloden, Papamoa
  - Lakeland Clinicaltrials Rotorua, Rotorua
  - Lakeland Clinicaltrials Wellington, Upper Hutt
- Philippines (3):
  - San Francisco Multi-Purpose Building, Manila
  - University of the East-Ramon Magsaysay Memorial Medical Center Inc., Manila
  - Health Index Multispeciality Clinic, Quezon City
- South Korea (16):
  - Korea University Ansan Hostpital, Ansan, Gyeonggi-do
  - Ajou university hospital, Suwon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha university hospital, Incheon
  - Seoul national university hosptial, Seoul
  - Soonchunhyang university hospital, Seoul
  - Ewha womans university medical center, Seoul
  - Hallym university medical center, Seoul
  - Korea university Anam hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Seoul
  - Wonju severance christian hospital, Wŏnju
- Thailand (4):
  - Armed Forces Research Institute of Medical Sciences, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Sriganarind Hospital, Khon Kaen
- Ukraine (7):
  - Medical center "Preventclinic" LLC, Dniprodzerzhyns'k, Dnipropetrovs'k
  - Treatment and Diagnostic Center of LLC Treatment and Diagnostic Center Adonis Plus, Dnipro
  - Medical and Diagnostic Сеntег of Рrivatе Еntеrрrisе of Рrivatе Manufacturing Соmрапу Acinus, Kropyvnytskyi
  - Communal non-profit enterprise Kyiv City Clinical Hospital №6, Kyiv
  - Medical Center "Ok!Clinic+" of International Institute of Clinical Research LLC, Kyiv
  - Municipal Nonprofit Enterprise "Khmelnytsky Regional Hospital for War Veterans" of Khmelnytsky Regional Council, Kyiv
  - Private Clinic LLC Blagomed, Odesa
- Pasteur Institute, Hochiminh City, Vietnam

REFERENCES:
- [Derived] Song JY, Choi WS, Heo JY, Kim EJ, Lee JS, Jung DS, Kim SW, Park KH, Eom JS, Jeong SJ, Lee J, Kwon KT, Choi HJ, Sohn JW, Kim YK, Yoo BW, Jang IJ, Capeding MZ, Roman F, Breuer T, Wysocki P, Carter L, Sahastrabuddhe S, Song M, D'Cor N, Kim H, Ryu JH, Lee SJ, Park YW, Cheong HJ; GBP510/AS03 study group. Immunogenicity and safety of SARS-CoV-2 recombinant protein nanoparticle vaccine GBP510 adjuvanted with AS03: interim results of a randomised, active-controlled, observer-blinded, phase 3 trial. EClinicalMedicine. 2023 Sep 7;64:102140. doi: 10.1016/j.eclinm.2023.102140. eCollection 2023 Oct. PMID 37711219
- [Derived] Walls AC, VanBlargan LA, Wu K, Choi A, Navarro MJ, Lee D, Avena L, Berrueta DM, Pham MN, Elbashir S, Kraft JC, Miranda MC, Kepl E, Johnson M, Blackstone A, Sprouse K, Fiala B, O'Connor MA, Brunette N, Arunachalam PS, Shirreff L, Rogers K, Carter L, Fuller DH, Villinger F, Pulendran B, Diamond MS, Edwards DK, King NP, Veesler D. Distinct sensitivities to SARS-CoV-2 variants in vaccinated humans and mice. Cell Rep. 2022 Aug 30;40(9):111299. doi: 10.1016/j.celrep.2022.111299. Epub 2022 Aug 15. PMID 35988541